CLINICAL TRIAL: NCT05480111
Title: The Role of Quadratus Lumborum Blocks Following Minimally Invasive Hysterectomy: A Blinded, Randomized Controlled Trial
Brief Title: The Role of Quadratus Lumborum Blocks Following Minimally Invasive Hysterectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Randa Jalloul, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HSC-MS-22-0158
Record Dates: First submitted 2022-06-28; First posted 2022-07-29 (Actual); Results first posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Pain, Postoperative
Keywords: laparoscopy; hysterectomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- QL Block (Experimental)
  Interventions: Drug: Sham Local; Drug: QL
- Local Anesthesia at incision site (Active Comparator)
  Interventions: Drug: Local anesthesia at incision site; Drug: Sham QL

INTERVENTIONS:
Drug: Local anesthesia at incision site — 20 ml of 0.25% Bupivacaine will be given at incision site
  Arms: Local Anesthesia at incision site
Drug: Sham QL — 20 mls of normal saline given at QL.The QL block will be administered on both the right and left sides. The transducer is placed transverse immediately cranial to the iliac crest and at the level of the posterior axillary line. The needle is then inserted inplane from the lateral edge of the transducer and advanced through the quadratus lumborum (QL) muscle until the needle tip penetrated the epimysium of the anterior part of the QL muscle. The anesthetic is injected after repeated negative aspiration tests for blood in the fascial interspace between the QL and psoas major (PM) muscles posterior to the transversalis fascia
  Arms: Local Anesthesia at incision site
Drug: Sham Local — 20 mls of normal saline given at incision site
  Arms: QL Block
Drug: QL — QL block involves injection of 19 ml of 0.25% Bupivacaine and iml(4mg) of Decadron in a fascial place formed partly by the posterior surface of the quadratus lumborum muscle.The QL block will be administered on both the right and left sides. The transducer is placed transverse immediately cranial to the iliac crest and at the level of the posterior axillary line. The needle is then inserted inplane from the lateral edge of the transducer and advanced through the quadratus lumborum (QL) muscle until the needle tip penetrated the epimysium of the anterior part of the QL muscle. The anesthetic is injected after repeated negative aspiration tests for blood in the fascial interspace between the QL and psoas major (PM) muscles posterior to the transversalis fascia
  Arms: QL Block

SUMMARY:
The purpose of this study is to compare quality of recovery as well as peri-operative systemic opiates use and pain scores in patients undergoing laparoscopic or robotic hysterectomy when local anesthetic versus Quadratus Lumborum nerve block (QL-2) is added to the standard pain management.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking
* American Society of Anesthesiologists (ASA) physical status 1-3
* Planned laparoscopic or robotic hysterectomy

Exclusion Criteria:

* History of chronic pain requiring preoperative opioids, Known alcoholism disorder
* Congenital coagulopathy,
* Localized soft tissue infection,
* Use of anticoagulants,
* Dementia, inability or refusal to provide consent for the surgery
* Morbid obesity (BMI > 50), due to expected technical difficulty to achieve the block

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randa J Jalloul, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | QL Block | Local Anesthesia at Incision Site
Started | 38 | 38
Follow up at 24 Hours | 32 | 37
Follow up at 6 Weeks | 29 | 34
Completed | 29 | 34
Not Completed | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Local Anesthesia at Incision Site | QL Block | Total
Number analyzed (Participants) | 38 | 38 | 76
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 44 [34 to 59] | 45 [35 to 57] | 44 [39 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 38 | 76
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 14 | 13 | 27
  Black or African American | 21 | 15 | 36
  Other/Unknown/Not Reported | 3 | 10 | 13
Region of Enrollment [Number; unit: participants]
  United States | 38 | 38 | 76
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 30 [23 to 42] | 35 [21 to 46] | 32.8 [26.5 to 38.5]
Number of Participants who are Nulliparous [Count of Participants; unit: Participants] | 10 | 8 | 18
Indication for the surgery [Count of Participants; unit: Participants]
  Symptomatic fibroids | 25 | 22 | 47
  Other (adenomyosis, polys, abnormal bleeding) | 13 | 16 | 29
History of Previous Uterine Surgery [Count of Participants; unit: Participants] — History of previous uterine Surgery, such as myomectomy or cesarean sections
  Participants | 29 | 33 | 62
American Society of Anesthesiology (ASA) Classification [Count of Participants; unit: Participants] — ASA Physical Status Classification System - The purpose of the system is to assess and communicate a patient's pre-anesthesia medical co-morbidities.
  ASA I :A normal healthy patient ASA II :A patient with mild systemic disease ASA III: A patient with severe systemic disease ASA IV: A patient with severe systemic disease that is a constant threat to life ASA V: A moribund patient who is not expected to survive without the operation ASA VI: A declared brain-dead patient whose organs are being removed for donor purposes
  Participants
    ASA I :A normal healthy patient | 21 | 21 | 42
    ASA II :A patient with mild systemic disease | 17 | 17 | 34
    ASA III: A patient with severe systemic disease | 0 | 0 | 0
    ASA IV: A patient with severe systemic disease that is a constant threat to life | 0 | 0 | 0
    ASA V: A moribund patient who is not expected to survive without the operation | 0 | 0 | 0
    ASA VI: A declared brain-dead patient whose organs are being removed for donor purposes | 0 | 0 | 0
Surgery Type [Count of Participants; unit: Participants]
  Robotic | 34 | 34 | 68
  Laparoscopic | 4 | 3 | 7
  Conversion to Open | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Pain as Assessed by the Quality of Recovery (QOR-40) Validated Questionnaire
Description: The QOR-40 questionnaire has 7 questions assessing pain with a maximum score of 35 and a minimum score of 5, a lower score indicating greater pain.
Time Frame: 24 hours after anesthesia
Population: Data was not collected for 1 participant in the Local Anesthesia at incision site arm. Data was not collected for 6 participants in the QL block arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Local Anesthesia at Incision Site | QL Block
Number analyzed (Participants) | 37 | 32
score on a scale | 30.0 (2.8) | 31.1 (2.2)

2. Primary Outcome: Physical Comfort as Assessed by the Quality of Recovery (QOR-40) Validated Questionnaire
Description: The QOR-40 questionnaire has 12 questions assessing physical comfort with a maximum score of 60 and a minimum score of 12, a lower score indicating a worst outcome.
Time Frame: 24 hours after anesthesia
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Local Anesthesia at Incision Site | QL Block
Number analyzed (Participants) | 37 | 32
score on a scale | 52.9 (4.9) | 54.3 (5.1)

3. Primary Outcome: Physical Independence as Assessed by the Quality of Recovery (QOR-40) Validated Questionnaire
Description: The QOR-40 questionnaire has 5 questions assessing physical independence, with a maximum score of 25 and a minimum score of 5, with a lower score indicating a worst outcome.
Time Frame: 24 hours after anesthesia
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Local Anesthesia at Incision Site | QL Block
Number analyzed (Participants) | 37 | 32
score on a scale | 20.4 (3.0) | 21.3 (2.4)

4. Primary Outcome: Psychological Support as Assessed by the Quality of Recovery (QOR-40) Validated Questionnaire
Description: The QOR-40 questionnaire has 7 questions assessing Psychological support, with a maximum score of 35 and a minimum score of 7, with a lower score indicating a worst outcome.
Time Frame: 24 hours after anesthesia
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Local Anesthesia at Incision Site | QL Block
Number analyzed (Participants) | 37 | 32
score on a scale | 30.2 (2.8) | 30.3 (1.7)

5. Primary Outcome: Emotional State as Assessed by the Quality of Recovery (QOR-40) Validated Questionnaire
Description: The QOR-40 questionnaire has 9 questions assessing emotional state, with a maximum score of 45 and a minimum score of 9, with a lower number indicating a worst outcome.
Time Frame: 24 hours after anesthesia
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Local Anesthesia at Incision Site | QL Block
Number analyzed (Participants) | 37 | 32
score on a scale | 42.2 (2.7) | 42.1 (4.0)

6. Primary Outcome: Quality of Recovery as Assessed by the Quality of Recovery (QOR-40) Validated Questionnaire
Description: The QOR-40 questionnaire has 40 questions with a total score from 40 (poorest quality of recovery) to 200 (best quality of recovery), with a higher score indicating a better outcome
Time Frame: 24 hours after anesthesia
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Local Anesthesia at Incision Site | QL Block
Number analyzed (Participants) | 37 | 32
score on a scale | 175.6 (9.7) | 179.1 (10.3)

7. Secondary Outcome: Pain at Rest as Assessed by the Visual Analog Scale
Description: 0 corresponding to no pain at all and 10 corresponding to worst imaginable pain
Time Frame: Post anesthesia care unit (PACU) immediately postoperatively
Population: Data was not collected for 1 participant in the Local Anesthesia at incision site arm. Data was not collected for 3 participants in the QL block arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Local Anesthesia at Incision Site | QL Block
Number analyzed (Participants) | 37 | 35
score on a scale | 2.2 (3.6) | 2.4 (3.8)

8. Secondary Outcome: Pain at Rest as Assessed by the Visual Analog Scale
Description: 0 corresponding to no pain at all and 10 corresponding to worst imaginable pain
Time Frame: At the time of first opiate administration(upto one day after surgery)
Population: Data was not collected for 3 participants in the Local Anesthesia at incision site arm. Data was not collected for 3 participants in the QL block arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Local Anesthesia at Incision Site | QL Block
Number analyzed (Participants) | 35 | 35
score on a scale | 7.6 (1.7) | 7.4 (2)

9. Secondary Outcome: Pain at Rest as Assessed by the Visual Analog Scale
Description: 0 corresponding to no pain at all and 10 corresponding to worst imaginable pain
Time Frame: At the time of discharge (upto 3 days after surgery)
Population: Data was not collected for 7 participants in the Local Anesthesia at incision site arm. Data was not collected for 9 participants in the QL block arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Local Anesthesia at Incision Site | QL Block
Number analyzed (Participants) | 31 | 29
score on a scale | 1.4 (1.8) | 1.3 (1.9)

10. Secondary Outcome: Pain at Rest as Assessed by the Visual Analog Scale
Description: 0 corresponding to no pain at all and 10 corresponding to worst imaginable pain
Time Frame: Day 1 (24+/=4 hours post surgery)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Local Anesthesia at Incision Site | QL Block
Number analyzed (Participants) | 37 | 32
score on a scale | 4.5 (2.2) | 4.5 (2.6)

11. Secondary Outcome: Pain at Dynamic as Assessed by the Visual Analog Scale
Description: 0 corresponding to no pain at all and 10 corresponding to worst imaginable pain
Time Frame: Day 1 (24+/=4 hours post surgery)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Local Anesthesia at Incision Site | QL Block
Number analyzed (Participants) | 37 | 32
score on a scale | 6.9 (2.2) | 6.7 (2.5)

12. Secondary Outcome: Pain at Rest as Assessed by the Visual Analog Scale
Description: 0 corresponding to no pain at all and 10 corresponding to worst imaginable pain
Time Frame: Day 14 post surgery
Population: Data was not collected for 2 participants in the Local Anesthesia at incision site arm. Data was not collected for 7 participants in the QL block arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Local Anesthesia at Incision Site | QL Block
Number analyzed (Participants) | 36 | 31
score on a scale | 2 (1.9) | 1.8 (2)

13. Secondary Outcome: Pain at Dynamic as Assessed by the Visual Analog Scale
Description: 0 corresponding to no pain at all and 10 corresponding to worst imaginable pain
Time Frame: Day 14 post surgery
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Local Anesthesia at Incision Site | QL Block
Number analyzed (Participants) | 36 | 31
score on a scale | 3.4 (2.2) | 3 (2.5)

14. Secondary Outcome: Pain at Rest as Assessed by the Visual Analog Scale
Description: 0 corresponding to no pain at all and 10 corresponding to worst imaginable pain
Time Frame: 6 weeks post surgery
Population: Data were not collected for 9 participants in the Local Anesthesia at incision site arm. Data were not collected for 4 participants in the QL Block arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Local Anesthesia at Incision Site | QL Block
Number analyzed (Participants) | 29 | 34
score on a scale | 0 (1) | 1 (2)

15. Secondary Outcome: Pain at Dynamic as Assessed by the Visual Analog Scale
Description: 0 corresponding to no pain at all and 10 corresponding to worst imaginable pain
Time Frame: 6 weeks post surgery
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Local Anesthesia at Incision Site | QL Block
Number analyzed (Participants) | 29 | 34
score on a scale | 0.8 (1.5) | 1 (1.8)

16. Secondary Outcome: Amount of Oral Morphine Consumed Measured in Morphine Milliequivalents (OME)
Time Frame: in PACU(upto 8 hours after surgery)
Population: Data was not collected for 3 participants in the Local Anesthesia at incision site arm. Data was not collected for 4 participants in the QL block arm.
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Local Anesthesia at Incision Site | QL Block
Number analyzed (Participants) | 35 | 34
milligrams | 9.77 (5.3) | 13.5 (19)

17. Secondary Outcome: Amount of Oral Morphine Consumed Measured in Morphine Milliequivalents (OME)
Time Frame: 24 hours after surgery
Population: Data was not collected for 3 participants in the Local Anesthesia at incision site arm. Data was not collected for 5 participants in the QL block arm.
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Local Anesthesia at Incision Site | QL Block
Number analyzed (Participants) | 35 | 33
milligrams | 36.48 (25) | 36.57 (24.8)

18. Secondary Outcome: Amount of Oral Morphine Consumed Measured in Morphine Milliequivalents (OME)
Time Frame: 2 weeks post surgery
Population: Data was not collected for 3 participants in the Local Anesthesia at incision site arm. Data was not collected for 6 participants in the QL block arm.
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Local Anesthesia at Incision Site | QL Block
Number analyzed (Participants) | 35 | 32
milligrams | 58.2 (43.9) | 60.69 (58.7)

19. Secondary Outcome: Amount of Oral Morphine Consumed Measured in Morphine Milliequivalents (OME)
Time Frame: 6 weeks post surgery
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Local Anesthesia at Incision Site | QL Block
Number analyzed (Participants) | 35 | 32
milligrams | 58.2 (43.9) | 60.69 (58.7)

20. Secondary Outcome: Time to Administration of First Pain Medication in PACU
Time Frame: From entry to Post anesthesia care unit (PACU) to time to administration of first pain medication in PACU (about 75 minutes)
Population: Data were not collected for 1 participant in the QL block
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Local Anesthesia at Incision Site | QL Block
Number analyzed (Participants) | 38 | 37
minutes | 63.3 (49) | 88.7 (85)

21. Secondary Outcome: Number of Participants With Complications Related to a Study Intervention
Time Frame: 30 days
Population: Data were not collected for 1 participant in the QL block arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Local Anesthesia at Incision Site | QL Block
Number analyzed (Participants) | 38 | 37
Participants | 0 | 0

22. Secondary Outcome: Postoperative Nausea and Vomiting (PONV) Score Before Discharge
Description: Postoperative Nausea and Vomiting (PONV) score before discharge
  Scale: (none, mild, moderate)
Time Frame: about 24 hours
Population: Data were not collected for 3 participants in the QL block arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Local Anesthesia at Incision Site | QL Block
Number analyzed (Participants) | 38 | 35
Participants
  None | 27 | 24
  Mild | 8 | 9
  Moderate | 3 | 2

23. Secondary Outcome: Time Needed to Administer the Intervention QL Block
Time Frame: Time to administration of intervention QL block
Population: Data were not collected for this outcome measure
Arm/Group | Local Anesthesia at Incision Site | QL Block
Number analyzed (Participants) | 0 | 0

24. Other Pre Specified Outcome: Number of Participants That Required Morcellation
Time Frame: Intraoperative (about 3 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Local Anesthesia at Incision Site | QL Block
Number analyzed (Participants) | 38 | 38
Participants
  Umbilical extraction site | 9 | 7
  Mini Laparotomy extraction site | 3 | 2
  Vaginal extraction site | 8 | 4

25. Other Pre Specified Outcome: Specimen Weight
Time Frame: inoperative (about 3 hours)
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Local Anesthesia at Incision Site | QL Block
Number analyzed (Participants) | 38 | 38
grams | 414.1 (521) | 297 (266)

26. Other Pre Specified Outcome: Duration of Surgery
Time Frame: about 3 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Local Anesthesia at Incision Site | QL Block
Number analyzed (Participants) | 38 | 38
minutes | 176 (62) | 178 (58)

27. Other Pre Specified Outcome: Number of Participants That Were Discharge on the Same Day
Time Frame: Hospital discharge (up to 24 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Local Anesthesia at Incision Site | QL Block
Number analyzed (Participants) | 38 | 38
Participants | 30 | 28

28. Other Pre Specified Outcome: Number of Participants for Which Lysis of Adhesions Took Greater Than 30 Minutes
Time Frame: about 3 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Local Anesthesia at Incision Site | QL Block
Number analyzed (Participants) | 38 | 38
Participants | 10 | 12

29. Other Pre Specified Outcome: Number of Participants With Intraoperative Complications
Time Frame: Intraoperative (about 3 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Local Anesthesia at Incision Site | QL Block
Number analyzed (Participants) | 38 | 38
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: 6 weeks post surgery
Arm/Group | QL Block | Local Anesthesia at Incision Site
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 12/38 | 14/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QL Block (N=38) | Local Anesthesia at Incision Site (N=38)
Cystotomy (Surgical and medical procedures) | 1 | 0
Cuff Cellulitis (Skin and subcutaneous tissue disorders) | 0 | 3
Nausea (General disorders) | 11 | 11
Vomiting (General disorders) | 11 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-18): https://cdn.clinicaltrials.gov/large-docs/11/NCT05480111/Prot_SAP_000.pdf